| IIDAD STUDY VISIT 1 | | | | | D | D | М | M | Υ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | CASE | REPO | RT FO | RM | | | | | |
| Prevalence of | Polycy | ystic ( | Ovary | Syn | drom | e in T | rinida | ad an | d To | ba |
| Study reference number: | | | | CRE | EC-SA.17 | 723/08/2 | 022 | | | |
| INSTITUTION: | | | | The Uni | versity o | f the We | est Indies | | | |
| | Door | C D:1. | <b>A</b> 1 | Mr. C. 1 | 044 | D. V. | 1 | 71 | D D | ·• |
| PRINCIPAL INVESTIGATOR: | Proi | f. Ricardo | | | | | Katesan S<br>Iohamme | | m, Dr. B | rian |
| I am confident that the information study was conducted in accordance | | | | | | | | | | |
| sinuy was commercia in accordance | | tained pr | | | | | | men m | ormen c | .0165 |
| Investigator's Signature: | | | | | | | 7 | | | |
| Date of signature: | | | | | | | | | | |
| | D D | M | M Y | Y | Y Y | | | | | |
| | MINIMU | UM REQ | UIRED | INFOR | RMATIO | N 1 | | | | |
| 1. Date of visit: | \ F | 178. 7 | | r A | T | | | A | | ÷ |
| 1. Date of visit: | | D | M M | V | V / | Y Y | ЭK | A | H | ı |
| | D | | IVI IVI | ( / ( ) | J | | 11 | <i>X</i> <b>X</b> | | 1 |
| 2. Age at first visit: | | | Y | r | [ | ☐ Don' | t know | | | |
| 3. Height ( <u>self-reported</u> ): | | | C: | m | [ | Don' | t know | | | |
| 4. Weight ( <u>self-reported</u> ): | | | K | g | [ | ☐ Don' | t know | | | |
| 5. What is the highest level of | Г | ] No Ed | luc | | | | | | | |
| education you have completed? | | ] Prima | | | | | | | | |
| | | Secon | • | | | | | | | • |
| | L | Tertia | ry<br>vocation | .a1 | | | | | | |
| 6. Is participant currently working | ·:? | - | complete | | | | No (w | hv) | | |
| | , | 001011 | elow | | | | | | | |
| 7. Occupation 1 - | Manageri | ial | | | □ 6 | – Self-l | Employed | d Farmin | ng | |
| | Technicia | ans and P | rofessior | nals | | - | oyee Farr | _ | | |
| <u> </u> | | | | | | | | | | |
| 3 - | Clerical/s<br>Services | secretary | | | | | d manual<br>lled man | | | |

**COMPLETED BY:** 

**SIGNATURE:** 

| SUBJECT ID: | | SU | BJECT | INITIA | LS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TDINI | DINIDAD CTUDY VICIT 4 | | | | | <b>D</b> | _ | B.4 | N/I | V | V |

| | CONTACT INFORMATION |
|---------------------------------------------|------------------------------|
| 1. Street address house number | |
| | Other district zone |
| 3. How long been living there? | years |
| 4. Telephone numbers (including area code): | Cell Home |
| 5.E-mail: NFID | Work HALL @RAFT |
| 6. Emergency contact: | Name: |
| | Relationship to participant: |
| | Telephone number 1: |
| | Telephone number 2: |

| | SUBJECT ID: | BJECT | INITIA | LS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| TRINI | TRINIDAD STUDY VISIT 1 | | | • | D | D | М | М | Υ | Υ |

| SOC | CIO - DI | EMOGRAPHIC INFORMA | TIO | N 1 |
|---|---|---|---|---|
| 1. Date of birth | | M M Y Y | | |
| 2. Ethnic Group (see below): | | Patient | | |
| Ethnicity group codes: | 1<br>2<br>3<br>4<br>5 | East Indian African Asian Mixed Other | | |
| 3. Religion: | | Anglican Catholic Methodist Presbyterian Pentecostal/Charismatic | | Other Christian Other Islam Traditional/Spiritualist Hindu No Religion |
| 4. Current marital status? | | Single Married Cohabitation Would rather not say | | Separated Divorced Widowed |
| 5. Participant's monthly income (in TT)? | | CATEGORY<br>Under 5,000<br>5,000 – 10,000<br>10,000 – 15,000 | | $15,000 - 20,000$ $20,000 - 25,000$ $\geq 26,000$ |

| SUBJECT ID: | SUBJECT INITIALS: | | VISIT DATE: | | | |
|---|---|---|---|---|---|---|
| TRINIDAD STUDY VISIT 1 | | D | D | M | M | Y |
| S | OCIO - DEMOGRAPHIC INFORMATI | ON 2 | | | | |
| 11. Has the participant ever smok or used tobacco products? | | | | No | | |
| S | OCIO - DEMOGRAPHIC INFORMATI | ION 3 | | | | |
| 12. Does the participant consume alcohol? | ☐ Yes ( <u>complete below</u> ) | | No ( <u>s</u> | <u>go to 14</u> ) | | |
| 13. Does the participant consume recreational drugs? | ☐ None ☐ Occasionally ☐ Specify | , [ | Daily<br>_ | , | | |
| S | OCIO - DEMOGRAPHIC INFORMATI | ION 4 | | | | |
| 14. How many minutes does the participant usually walk outside home every day? | less than 10 minutes 10-19 minutes 20-39 minutes 40-59 minutes ≥1 hour | | R | A | F | Γ |
| 15. How often does the subject do exercises? (works up a sweat with increased heart rate: aerobic, jogging, tennis, swimming) | ☐ 1 day per week ☐ 2 days per week ☐ 3 days per week ☐ 4 days per week ☐ ≥5 days per week | | ] Non | e | | |
| 16. How strenuous is the subject's exercise? | Mild (slow dancing, bowling, golf) Moderate (not exhausting: biking, Strenuous (sweats and increased he | treadmill, | | | y) tennis, | |

| | SUBJECT ID: | SU | BJECT | INITIA | LS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TRINIDAD STUDY VISIT 1 | | | | | • | D | D | М | М | Υ | Υ |

| | ME | DICAL HISTORY 1 |
|---|---|---|
| Please | check if the participant has had any of the foll | owing conditions in the past, or at present |
| | Cardiac High Blood Pressure Heart Attack Heart Murmur Irregular Heartbeat Mitral Valve Prolapse Peripheral Vascular Disease Stroke Other | 2 Endocrine Diabetes/sugar problems Thyroid disease Bone loss High Cholesterol Steroid Use Other |
| 3 | Respiratory Asthma Chronic Cough Bronchitis Emphysema Other | 4 Neurologic Spine/Back Injury Multiple Sclerosis Parkinson's Stroke Seizure Disorder/Epilepsy Other |
| 50000000 | Gastrointestinal Stomach Ulcers Irritable Bowel Constipation Diverticulitis Ulcerative colitis Crohn's Disease Other | 6 Bleeding Disorders Chronic Aspirin Use History of Blood Clot Platelet Problem Blood Transfusion Other |
| 7 | Genito-Urinary/Reproductive Recurrent urine infections Kidney stones Difficulty getting pregnant Menopausal symptoms Other | 8 Cancer Breast Cancer Lung Cancer Ovarian Cancer Thyroid Cancer Uterine Cancer Cervical Cancer Colon Cancer |
| 9 | Musculo-skeletal | 10 Sleep Disturbance Difficulty falling asleep Mulitiple episodes of waking at night Excessive sleepiness during the day Other (snoring) (sleep ap form) |

| SUBJECT ID: | SU | BJECT INITIALS: | | | VISI | T DAT | <b>E</b> : | |
|---|---|---|---|---|---|---|---|---|
| TRINIDAD STUDY VISIT 1 | | | D | D | M | M | Y | <u> </u> |
| | | 11 Other | | | | | | |
| | N | MEDICAL HISTORY 2 | 2 | | | | | |
| 10. What has been the participant's | | (Mark only one) | | | | | | |
| weight change during adult life (do not include times of pregnancy or | | Weight has stayed about the same (within 5 kg) | | | | | | |
| sickness)? How much? | | Steady weight gain | | | | | | |
| | | Lost weight as an adul | lt and kept | it off | | | | |
| | | Weight has gone up an | nd down n | nore than | 5 kg. | | | |
| 11. Is the participant on any special diet? | | Yes Specify | | | □ No | | | |

# CONFIDENTIAL DRAFT

| | SI | JBJEC | T ID: | | SL | LS: | | | | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TRIN | IDAD S | TUDY \ | /ISIT 1 | | | | | | | ) | D | M | M | Y | ` |
| | | | | | | ГORY | | | | | | | | | |
| | participa<br>ectomy? | ant had a | a | | | aplete be | | roki | | | No ( <u>go</u> | o to 2) | | | |
| | | | | | Uterus<br>Uterus + | 1 ovary | | | | | Uterus | s + both o | ovaries | | |
| | | | | Date Detail | M M | I M | Y YM | [ | | | | | | | |
| other | s particip<br>surgeries<br>tric. remo | (lapros | copy, | | Yes ( <u>con</u> | aplete be | llow) | | | | No | | | | |
| | | ] | List other | · surgerio | | gone, the<br>luding do | | | ere it w | as pe | rforme | d, | | | |
| 1 | | | | | | | | | | | | | | | |
| 2 | 0] | VI | | H | | | IA | M | M | Y | Y | A | F | | |
| | | | | | | | | M | M | Y | Y | | | | |
| 3 | | | | | | | | | | | | | | | |
| | | | | | | | | M | M | Y | Y | | | | |
| 4 | | | | | | | | M | M | Y | Y | | | | |
| 5 | | | | | | | | M | M | Y | Y | | | | |

No

Yes

Continued, see attached

| | SUBJECT ID: | SUBJECT | INITIALS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| TRIN | NIDAD STUDY VISIT 1 | 1 | | D | D | М | М | Υ | Υ |
| | | MEDIO | CATIONS | | | | | | |
| previ<br>horm | participant currently or iously taking any onnal contraceptive or ormin? | Yes (complete | e below) | | | No | | | |
| | Name | No. of years used | Start Date (MM/YY) | | Stop Da<br>(MM/Y) | | Sti | ll taking | |
| | OCP "" | | | | | | | | |
| | Estrogens "" | | | | | | | | |
| | Vaginal ring | | | | | | | | |
| | Transdermal patch | | | | | | | | |
| | Mirena IUD | | | | | | | | |
| | Transdermal Implant | | | | | | | | |
| | Injectable contraceptive | | | | | | | | |
| | Metformin ( mg/day) | | | | | | | | |
| | Infertility medications | | | | | | | | |
| | Others | | | | | | | | |
| | her medications, incl. nins & herbals? | Yes (list medi | cations below) | | R | No | | T | |
| | Medication and name | Dose | Start Date (MM/YY) | | Stop Da<br><i>(MM/Y)</i> | | Sti | ll taking | |
| 1 | | | | | | | | | |
| 2 | | | | | | | | | |
| 3 | | | | | | | | | |
| 4 | | | | | | | | | |
| 5 | | | | | | | | | |
| Cont | inued, see attached | | | П | No | u. | | | |

| SUBJECT ID: | | SU | BJECT | INITIA | LS: | | : | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TRINI | TRINIDAD STUDY VISIT 1 | | | | | D | D | М | М | Υ | Υ |

| | GYNECOLOGIC HISTORY 1 |
|---|---|
| 1. Age at 1st period? | Years |
| 2. The subject's periods are: | Regular Have stopped Irregular (complete 5 & 6) Never started |
| 3. What is/was the average length of menstrual cycles? | Days* (place a note) |
| *Days | between the start of one period and the start of the next |
| 4. What is/was the average No. menses cycles per year? | |
| 5. Date of last menstrual period: | D D M M Y Y |
| CONFI | DENTIAL DRAFT |

| SUBJECT ID: | SU | BJECT INITIAL | S: | | VISIT | DATE | : | |
|---|---|---|---|---|---|---|---|---|
| TRINIDAD STUDY VISIT 1 | | | D | D | M | M | Υ | Y |
| TRINIDAD GTODT VIOLET | | | | | 141 | 141 | • | • |
| GY | NEC | OLOGIC HISTO | RY 2 | | | | | |
| 5. Is the participant in menopause? | Ш | Yes (complete b | | | ☐ No | | | |
| | | Natural meno | opause | | | | | |
| | | Surgical men | opause | | | | | |
| 6. Does the participant have any | | Yes (complete b | elow) | | ☐ No | | | |
| menopausal symptoms? Which? | | | | | | | | |
| | | Hot flashes | | | | | | |
| | | Night sweats Other | | | | | | |
| | Ш | Other | | | | | | |
| 7. In total, how long has the participant been in menopause? | | Less than 1 year | | | 1-2 years | | | |
| ocen in menopulase. | | 2-4 years | | Ш | More than | 4 years | | |
| 9 H | | $\neg$ | | | | | | |
| 8. How old was participant when she stopped having periods? | | Years | | | | | | |
| CONFIDE | | | T | JI | $) \land$ | E | | |
| <del>UUNIIDE</del> | 1 | | | /1 | | | | |
| | YNE | COLOGIC REVI | EW 3 | | | | | |
| 9. Is the participant sexually active? | | Yes (complete b | oelow) | | No, never | had sex | | |
| | | No, but previou active (answer l | | | | | | |
| | | | , | | | | | |
| | | How long? | | | | | | |
| 10. Frequency of sex? | | More than 2 time | es a week | | | | | |
| | | Less than 2 time | s a week | | | | | |
| | | | | - | | | | 1 |
| 11. Has the participant ever tried to | | Yes (go to 13) | | | No (go to | 24) | | |
| become pregnant for more than 1 year, with no success? | | Don't know (go | to 13) | | 110 ( <u>20 10</u> | <u>~</u> ") | | |
| with no success? | | 2011 t Know ( <u>20</u> | <u></u> j | | | | | |
| 12. Did the participant visit a doctor/clinic | | Yes (go to 13) | | | No (go to | 24) | | |
| because of infertility? | _ | ( <u>=</u> / | | | \ <u>=</u> | | | |

| SUBJECT ID: | SU | BJEC1 | INITIA | LS: | | | VISI | T DATE | 3 |
|---|---|---|---|---|---|---|---|---|---|
| TRINIDAD STUDY VISIT 1 | | | | | D | D | M | M | Υ |
| 13. Was the reason for infertility found? | | Yes ( | <u>go to 14</u> ) | 1 | | □ N | o ( <u>go to</u> | <u>15</u> ) | |
| 14. What was the reason of infertility? | | Ovula | ation/mer | nstruation | problem | ı — | | | |
| | | Horm<br>PCOS | ional prol<br>S | blem | | | | es/uterus<br>ometrios | s problem<br>is |
| | | | e infectio<br>ature mer | | | | | olem witl<br>er age | h partner |
| | | | | _ | | | | 't know | |
| | | Other<br>Speci | problem | | | | | | |
| | CVNE | COLOG | SIC REV | TEW 4 | | _ | | | |
| 15.15 | GINE | COLOG | JIC KEV | TEW 4 | | | | | |
| 15. How many pregnancies did the participant have? | | | | | | | | | |
| 16. How old was the | | | | | | | | | |
| participant at the end of her <u>first</u> pregnancy? | years | | TA | <b>XL</b> | T | )R | Δ | F | Τ |
| 17. How old was the | <b>1</b> | 1 | 11 | | | /1/ | <u> </u> | | 1 |
| participant at the end of her last pregnancy? | years | S | | | | | | | |
| 18. № of live birth(s) | | | | | | | | | |
| | <u> </u> | | | | | | | | |
| 19. № of stillbirth(s) | | | | | | | | | |
| 20. № of ectopic pregnancies | | | | | | | | | |
| | <b>_</b> | | | | | | | | |
| 21. № of miscarriages | | | | | | | | | |
| 22. № of elective/induced abortion(s) | | | | | | | | | |

| | SI | JBJEC | T ID: | | SU | BJECT | INITIA | LS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TDINI | DVD 6. | TUDV | /ICIT 4 | • | | | | | <u> </u> | <u> </u> | RA | RA | V | v |

| | GYNECOLOGIC REVIEW 5 | |
|---|---|---|
| 23. Does the participant complain of acne? | Yes (complete below) | No |
| | Age first noticed: years | |
| 24. Does the participant complain of scalp hair loss? | ☐ Yes ( <u>complete below</u> ) | No No |
| | Age first noticed: years | |
| 25. In the below figure have participant mark how much scalp hair loss she has had. | | |



| | SI | JBJEC | T ID: | | SU | BJECT | INITIA | LS: | VISIT DATE: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TRINI | DAD S | TUDY \ | /ISIT 1 | • | | | | • | D | D | М | М | Υ | Υ |

| | | GYNECOLOGIC REVIEW 9 | |
|---|---|---|---|
| 26. Does the participant have excessive or unwanted hair | | Yes (complete below) | No |
| growth? | | Age first noticed | |
| 27. Does the participant remove excess body or facial | | Yes (complete below)* | No |
| hair (using electrolysis, lasers, shaving, creams, threading, | | Upper lip | Upper abdomen |
| etc.)? | | Chin | Lower abdomen |
| If yes, on what body part? | | Chest | Upper arms |
| | | Upper back | Thighs |
| | | Lower back | |
| | *Not | the lower legs or lower arms/forearms | |

## HYPERANDROGENIC FEATURES EVALUATION RECORD

## Modified Ferriman-Gallwey Hirsutism Score



Total modified F-G score:

| S | UBJEC <sup>*</sup> | T ID: | | SU | IBJEC1 | INITIA | LS: | | VISIT | DATE | : | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| GH-P | EP STI | JDY VI | SIT 1 | | | | 1 | <br>D | M | M | Υ | Y |

## BECKS INVENTORY 1

## 28. Please complete below:

| 1. | _ | _ |
|---|---|---|
| | 0 | I do not feel sad. |
| | ĭ | I feel sad |
| | _ | |
| | 2 | I am sad all the time and I can't snap out of it. |
| _ | 3 | I am so sad and unhappy that I can't stand it. |
| 2. | | |
| | 0 | I am not particularly discouraged about the future. |
| | 1 | I feel discouraged about the future. |
| | 2 | I feel I have nothing to look forward to. |
| | 3 | I feel the future is hopeless and that things cannot improve. |
| 3. | _ | |
| - | 0 | I do not feel like a failure. |
| | 1 | |
| | | I feel I have failed more than the average person. |
| | 2 | As I look back on my life, all I can see is a lot of failures. |
| _ | 3 | I feel I am a complete failure as a person. |
| 4. | | |
| | 0 | I get as much satisfaction out of things as I used to. |
| | 1 | I don't enjoy things the way I used to. |
| | 2 | I don't get real satisfaction out of anything anymore. |
| | 3 | I am dissatisfied or bored with everything. |
| 5. | | |
| | 0 | I don't feel particularly guilty |
| | ĭ | I feel guilty a good part of the time. |
| | 2 | |
| | 3 | I feel quite guilty most of the time. |
| _ | - 3 | I feel guilty all of the time. |
| 6. | | T1 60 1T 1 1 1 1 1 1 |
| | 0 | I don't feel I am being punished. |
| | 1 | I feel I may be punished. |
| | 2 | I expect to be punished. |
| | 3 | I feel I am being punished. |
| 7. | | |
| | 0 | I don't feel disappointed in myself. |
| | 1 | I am disappointed in myself. |
| | 2 | I am disgusted with myself. |
| | 3 | I hate myself. |
| 8. | | Thate my seit. |
| ٥. | 0 | I don't feel I am any worse than anybody else. |
| | i | |
| | | I am critical of myself for my weaknesses or mistakes. |
| | 2 | I blame myself all the time for my faults. |
| _ | 3 | I blame myself for everything bad that happens. |
| 9. | _ | |
| | 0 | I don't have any thoughts of killing myself. |
| | 1 | I have thoughts of killing myself, but I would not carry them out. |
| | 2 | I would like to kill myself. |
| | 3 | I would kill myself if I had the chance. |
| 10. | | , and the second |
| | 0 | I don't cry any more than usual. |
| | ĭ | I cry more now than I used to. |
| | 2 | I cry all the time now. |
| | 3 | I used to be able to cry, but now I can't cry even though I want to. |
| | _ | a more to be note to cay, but now a court cay even mough a wall to. |

#### **BECKS INVENTORY 2**

#### 29. Please complete below (cont.):

```
11.
               I am no more irritated by things than I ever was.
               I am slightly more irritated now than usual.
    1
                I am quite annoyed or irritated a good deal of the time.
    3
               I feel irritated all the time.
12.
     0
               I have not lost interest in other people.
               I am less interested in other people than I used to be.
                I have lost most of my interest in other people.
     3
               I have lost all of my interest in other people.
13.
     0
                I make decisions about as well as I ever could.
               I put off making decisions more than I used to.
               I have greater difficulty in making decisions more than I used to.
     2
     3
               I can't make decisions at all anymore.
14.
     0
               I don't feel that I look any worse than I used to.
               I am worried that I am looking old or unattractive.
     1
     2
               I feel there are permanent changes in my appearance that make me look
                unattractive
     3
               I believe that I look ugly.
15.
     0
               I can work about as well as before.
     1
               It takes an extra effort to get started at doing something.
     2
               I have to push myself very hard to do anything.
     3
               I can't do any work at all.
16.
     0
               I can sleep as well as usual.
               I don't sleep as well as I used to.
               I wake up 1-2 hours earlier than usual and find it hard to get back to sleep.
     2
     3
               I wake up several hours earlier than I used to and cannot get back to sleep.
17.
               I don't get more tired than usual.
    0
               I get tired more easily than I used to.
    1
    )
               I get tired from doing almost anything.
    3
               I am too tired to do anything.
18.
    0
               My appetite is no worse than usual.
    1
               My appetite is not as good as it used to be.
                My appetite is much worse now.
               I have no appetite at all anymore.
19.
    0
               I haven't lost much weight, if any, lately.
               I have lost more than five pounds.
    1
               I have lost more than ten pounds.
I have lost more than fifteen pounds.
    2
```

### **BECKS INVENTORY 3**

### 30. Please complete below (cont.):

| icase comp | nete below (cont.). |
|---|---|
| 20. | |
| 0 | I am no more worried about my health than usual. |
| 1 | I am worried about physical problems like aches, pains, upset stomach, or constipation. |
| 2 | I am very worried about physical problems and it's hard to think of much else. |
| 3 | I am so worried about my physical problems that I cannot think of anything else. |
| 21. | |
| 0 | I have not noticed any recent change in my interest in sex. |
| 1 | I am less interested in sex than I used to be. |
| 2 | I have almost no interest in sex. |
| 3 | I have lost interest in sex completely. |

| | | | SF-12 | | | | |
|---|---|---|---|---|---|---|---|
| 31. Please com | plete below (cont.) | ): | | | | | |
| l. In general, w | ould you say your | health is: | | | | | |
| □₁ Excellent | □₂ Very good | □₃ Good | □₄ Fair | | □s Poor | | |
| | questions are abou<br>se activities? If so | | might do duri | ng a typic | al day. Does | your health | low |
| | | | YES,<br>limited<br>a lot | | YES,<br>limited<br>a little | NO, no<br>limited<br>at all | |
| | ivities such as moving<br>eaner, bowling, or pla | | □1 | | □2 | □₃ | |
| | veral flights of stairs. | | <b>□</b> 1 | | □2 | | |
| | t 4 weeks, have yo | | | oblems wi | | or other rea | ular |
| | as a result of your | _ | | | , | | |
| | | | | YES | | NO | |
| 4. Accomplish | ned less than you w | ould like. | | D <sub>1</sub> | | □2 | |
| • | in the kind of work | | es. | D <sub>1</sub> | | <b>□</b> 2 | |
| | t 4 weeks, have yo | | | | th your work | | ular |
| | as a result of any | | | | | | |
| , | | | (3000) | | <b></b> | | |
| | | | | YES | | NO | |
| B. Accomplish | ed less than you wo | ould like. | | D <sub>1</sub> | | <b>□</b> 2 | |
| 7. Did work or a | ctivities less carefu | illy than usual. | | □ <sub>1</sub> | | <b>□</b> 2 | |
| | ast 4 weeks, how | - | | vour norm | al work (incl | udina work o | utside |
| the home and h | | | | | | <b>_</b> | |
| | • | | | | | | |
| □₁ Not at all | □₂ A little bit | □₃ Mod | derately | □₄ Quite | a bit | □s Extreme | ely |
| These question | ns are about how y | ou have been f | eeling during t | the past 4 | weeks. | | |
| | ion, please give th | | | | | ve been feeli | ng. |
| How much of the | he time during the | past 4 weeks | - | | | | |
| | | All of | Most | A good | Some | A little | |
| | | the | of the | bit of | of the | of the | of the |
| | -1-0 | time | time | the time | time | time | time |
| ). Have you felt o | • | □1 | □2 | □₃ | □4 | □s | □6 |
| 10. Did you have | | □1 | □2 | □s | □4 | □s | □6 |
| 11. Have you felt of blue? | down-hearted and | □1 | □2 | □₃ | □4 | □s | □6 |
| 12. During the | past 4 weeks, how | much of the ti | me has your p | hysical he | alth or emoti | onal problem | 15 |
| | your social activiti | | | | | | _ |
| | _ | | • | | | | |
| ☐₁ All of the tim | e □₂ Most of the t | ime 🗅 Sor | ne of the time | □₄ A littl | e of the time | □s None of | the time |

# RUTA MENORRGHIA SCALE 1

# 32. Please complete below: gyne history 1

| <ul> <li>1. On average, during the last three months, for how many days did your period last? (Please tick one box)</li> <li>Less than 3 days 0</li> <li>Between 3 and 7 days 0</li> <li>Between 8 and 10 days 0</li> </ul> |
|---|
| □ More than 10 days 0 |
| 2. On average, during the last three months, were your periods regular or irregular? (Please |
| tick one box) Regular |
| □ Irregular |
| 3. On average, during the last three months, how many days were there from the first day of a period to the first day of |
| the next period? (Please tick one box) |
| □ Less than 21 days |
| <ul> <li>Between 21 and 35 days</li> <li>More than 35 days</li> </ul> |
| a Word than 33 days |
| 4. On average, during the last three months, would you describe your periods as? (Please tick one box) |
| □ Light |
| □ Moderate |
| □ Heavy □ Very Heavy |
| STONE OF THE PRODUCTION OF |
| 5. On average, during the last three months, for how many days of each period was the bleeding heavy? (Please tick one |
| box) |
| □ Not heavy |
| □ Between 1 and 3 days |
| <ul> <li>□ Between 4 and 6 days</li> <li>□ Between 7 and 10 days</li> </ul> |
| □ More than 10 days |
| 6. During the last three months, have you passed any clots of blood? (Please tick one box) |
| □ Yes |
| □ No |
| 7. On average, during the last three months, have your periods been associated with any pain? (Please tick one box) |
| □ No pain at all |
| □ Slight pain |
| □ Moderate pain |
| <ul> <li>Severe pain</li> <li>Very severe pain</li> </ul> |
| u very severe parit |
| 8. On average, during the last three months, have you had any problems with soiling/staining any of the following because of |
| your periods? (Please tick one box) |
| □ Soiling/staining of your underclothes/undergarments |
| □ Soiling/staining of your outer clothes/over garments |
| <ul> <li>Soiling/staining of your bed linen</li> <li>Soiling/staining of your upholstery</li> </ul> |
| □ Soiling/staining of your upholstery |

| | RUTA MENORRGHIA SCALE 2 |
|---|---|
| 34. Please complete below (cont.): | |
| 9. On av | rerage, during the last three months, have your periods prevented you from carrying out your work, housework |
| or other daily activities? (Please tick one box) | |
| | No, not at all |
| | I could continue to work, but my work suffered |
| | Yes, usually with no more than one day with each period Yes, usually more than one day with each period |
| | res, askany more than one day with each period |
| 10. On a | verage, during the last three months, have you been confined to bed with each period? (Please tick |
| one box | |
| | No, not at all |
| | Yes, usually for part of one day |
| | Yes, usually for the whole of one day Yes, usually for more than one day |
| Ш | res, usually for filore trial one day |
| 11. On a | overage, during the last three months, have your leisure activities been affected by your heavy periods? |
| (includir | ng sport, hobbies, social life)(Please tick one box) |
| | Not affected by heavy periods |
| | Mildly affected by heavy periods |
| | Moderately affected by heavy periods |
| | Severely affected by heavy periods |
| | Heavy periods have prevented any social life at all |
| 12. On a | overage, during the last three months, has your sex life been affected by your heavy periods? (Please tick one box) |
| | Not affected by heavy periods |
| | Mildly affected by heavy periods |
| | Moderately affected by heavy periods |
| | Severely affected by heavy periods Heavy periods prevented any sex life at all |
| | Does not apply |
| | verage, during the last three months, how many tampons might you use on the heaviest day of your period? |
| HARL CHARACTERSON | tick one box) |
| | No tampons at all |
| | Between 1 and 5 tampons Between 6 and 10 tampons |
| | Between 11 and 15 tampons |
| | More than 15 tampons |
| 14. On a | verage, how many pads might you use on the heaviest day of your period? (Please tick one box) |
| | No pads at all |
| | Between 1 and 5 pads |
| | Between 6 and 10 pads Between 11 and 15 pads |
| | More than 15 pads |
| 1000 | And the second s |

15. At any time during the last three months, did you require more than one form of protection at the same time (Not including mini pads or mini pant-liners)? (Please tick one box)

| No |
|-----------------------------------------------------------------|
| Tampon and pad together |
| Two pads together |
| Tampon and two pads together |
| More protection than this (ie. disposable nappies, towels etc.) |

Weight

Height

Waist

Hip

# CONFIDENTIAL DRAFT